CLINICAL TRIAL: NCT07148401
Title: Parental and Patient Satisfaction of Hall Technique for Caries Management in Primary Molars
Brief Title: Parental Satisfaction of Hall Technique for Caries Management in Primary Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Lamia Mohamed Khairy Gadallah, Researcher, National Research Centre, Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18427
Record Dates: First submitted 2025-08-23; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hall technique (Active Comparator): stainless steel crown is inserted on indicated carious primary molars without tooth preparation
  Interventions: Device: Hall technique

INTERVENTIONS:
Device: Hall technique — Hall technique for placement of crowns on carious primary molars

SUMMARY:
As a newly introduced technique for caries management in primary teeth, patient-centered outcomes such as parental satisfaction, acceptability of the treatment and child discomfort needs to be investigated about Hall technique. Therefore , the aim of our study is to investigate parental and patient satisfaction of Hall technique in managing carious primary molars in children.

DETAILED DESCRIPTION:
Children included are those aged from 4 -10 years old. Children with one or more primary molar with class I and class II carious lesions, with no history of pain, or signs of reversible pulpitis .

Patients with signs of irreversible pulpitis as spontaneous pain or pain at night or pathological signs as periapical radiolucency and pathological root resorptions are excluded

Method:

Patient will receive no local anesthesia or tooth preparation. A proper sized preformed stainless-steel crown will be checked first. Then, the crown will be cemented on the tooth using glass ionomer cement The child is instructed to bite on the crown by means of a cotton roll. Excess cement was cleared immediately using a probe after cementation.

Primary outcome:

Parent satisfaction :

Parents satisfaction will be measured by a 5 point Likert scale with five possible answers: strongly agree, agree, neutral, disagree, and strongly disagree.[9]

Patient discomfort:

Discomfort at time of intervention: The Wong-Baker Faces Pain Scale will be used for assessment

Secondary outcomes:

Clinical evaluation will be performed at two-week interval, 6 and 12 months including :

Absence of adverse signs and symptoms of the carious lesion. Crown evaluation including crown retention.

ELIGIBILITY:
Inclusion Criteria:

* Children with one or more primary molar with class I and class II carious lesions.
* Teeth with no history of pain, or signs of reversible pulpitis

Exclusion Criteria:

* Teeth with signs of irreversible pulpitis as spontaneous pain or pain at night.
* Teeth with signs of non-vitality as presence of sinus or fistula or pathologic mobility.
* Teeth with pathological radiographic signs as periapical radiolucency and pathological root resorptions.
* Parental refusal for the use of stainless steel crown

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Parental satisfaction | at time of insertion, 2 weeks , 6 months, 1 year
  Parents satisfaction will be measured by a 5 point Likert scale with five possible answers: strongly agree, agree, neutral, disagree, and strongly disagree

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Centre, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
If scientific data with all required details are published so there will be no need to share individual participant data

REFERENCES:
- [Background] Hu S, BaniHani A, Nevitt S, Maden M, Santamaria RM, Albadri S. Hall technique for primary teeth: A systematic review and meta-analysis. Jpn Dent Sci Rev. 2022 Nov;58:286-297. doi: 10.1016/j.jdsr.2022.09.003. Epub 2022 Sep 27. PMID 36185501
- [Background] Innes NP, Evans DJ, Bonifacio CC, Geneser M, Hesse D, Heimer M, Kanellis M, Machiulskiene V, Narbutaite J, Olegario IC, Owais A, Araujo MP, Raggio DP, Splieth C, van Amerongen E, Weber-Gasparoni K, Santamaria RM. The Hall Technique 10 years on: Questions and answers. Br Dent J. 2017 Mar 24;222(6):478-483. doi: 10.1038/sj.bdj.2017.273. PMID 28336976
- [Background] Innes NP, Evans DJ. Modern approaches to caries management of the primary dentition. Br Dent J. 2013 Jun;214(11):559-66. doi: 10.1038/sj.bdj.2013.529. PMID 23744209